CLINICAL TRIAL: NCT00059800
Title: A Phase II Trial For Neutron Capture Therapy In Melanoma
Brief Title: Boron Neutron Capture Therapy in Treating Patients With Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Purpose: Treatment
Other Study IDs: BIDMC-W-01-0380-FB; CDR0000287207 (Registry Identifier: PDQ (Physician Data Query)); BIDMC-2001-P-001946
Record Dates: First submitted 2003-05-06; First posted 2003-05-07 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2005-12

CONDITIONS: Melanoma (Skin)
Keywords: recurrent melanoma; stage 0 melanoma; stage I melanoma; stage II melanoma; stage III melanoma; stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — Boron Neutron Capture Therapy

INTERVENTIONS:
Radiation: boron neutron capture therapy

SUMMARY:
RATIONALE: Boron neutron capture therapy may selectively kill tumor cells without harming normal tissue.

PURPOSE: Phase II trial to study the effectiveness of boron neutron capture therapy in treating patients who have melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the clinical response, by serial objective measurements, in patients with melanoma treated with boron neutron capture therapy.
* Determine the time course, uniformity, and severity of acute dermal reactions in patients treated with this regimen.
* Determine the late dermal reactions in patients who are followed for at least 6 months after treatment with this regimen.
* Determine the pharmacokinetics of this regimen in these patients.

OUTLINE: Patients are stratified according to tumor size (no greater than 15 cc vs greater than 15 cc).

Patients undergo boron neutron capture therapy.

Patients are followed for 3 years.

PROJECTED ACCRUAL: A total of 36 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed melanoma
* Evaluable disease
* Lesion(s) to be irradiated must be located in 1 of the following areas:

  * On an extremity
  * On the head or neck (including the scalp)
  * In the subdermal lymphatics (excluding the proximal axilla)
* Area to be irradiated must not exceed a maximum dimension of 10 cm

  * Maximum tumor depth from the surface of the skin cannot exceed 6 cm

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* More than 6 months

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Creatinine normal

Cardiovascular

* No history of severe cardiac disease
* No uncontrolled arrhythmias or conduction defects
* No unstable or newly diagnosed angina pectoris
* No recent coronary artery disease
* No congestive heart failure

Other

* Not pregnant
* Negative pregnancy test
* No history of phenylketonuria
* Must have sufficient mental competence

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy to study sites

Surgery

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-05; Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Clinical response
Time course, uniformity, and severity of acute dermal reactions
Late dermal reaction after at least six months
Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Paul M. Busse, MD, PhD, Study Chair — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Massachusetts Institute of Technology, Cambridge, Massachusetts